CLINICAL TRIAL: NCT04208282
Title: Safety and Efficacy of 7-day Wear Infusion Set vs. Control Infusion Set.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dr. Jacob Ilany MD, M.D., Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Arm A (Experimental): Quickset infusion system for the Phase 1. At day 28 or after using 4 sets , the patients will return to a visit, return all the extracted catheters sets and will switch to the 7 day set infusion set, entering Phase 2.
  Interventions: Device: 7 day infusion set
- Trial Arm B (Active Comparator): 7 day set infusion set for the Phase 1. At day 28 or after using 4 sets , the patients will return to a visit, return all the extracted catheters sets and will switch to the Quickset infusion systems , entering Phase 2.
  Interventions: Device: 7 day infusion set

INTERVENTIONS:
Device: 7 day infusion set — 7 days survival of the sets

SUMMARY:
The purpose of this study is to evaluate the Extended Wear (EW) infusion set seven day functioning in patients with Type 1 diabetes compared to the Quick-set infusion set. The study will be carried out in adults with type 1 diabetes.

DETAILED DESCRIPTION:
This is a 1-center, prospective, open label randomized, crossover controlled study.

40 patients will be using 4 infusion sets (a total of 160 sets) that will serve as an exploratory pilot study to assess the SD of 7 day use for future study design.

Eligible patients meeting the enrollment and randomization criteria will be randomized into 2 arms, each arm will undergo 2 phases. In each phase a different type of infusion set will be evaluated. Each evaluation will be for4 sets (up to 28 days). The order will be determined by the randomization process:

* Arm 1: Quick-EWIS. First phase Quickset, second phase EWIS.
* Arm 2: EWIS-Quick. First phase EWIS, second phase Quickset.

Following screening and informed consenting to the trial, a randomized procedure will define the subject trial arm:

* Trial Arm A: Subjects will be randomized to a group who will be using the Quickset infusion system for the Phase 1. All patients will be retrained on the use of the Quickset infusion set by site staff and will be asked to demonstrate proficiency. All subjects will be instructed to change sets every 7 days or at set failure (replace with another Quick-set). At day 28 or after using 4 sets (set used defined as a set that was used for more than 6 hours), the patients will return to a visit, return all the extracted catheters sets and will switch to the X infusion set, entering Phase 2. All patients will be trained at this visit on the use of the X EW infusion set by site staff and demonstrate proficiency in the use of the EW infusion set. After 28 days or after using 4 sets, the patients will return all the extracted catheters sets .
* Trial Arm B: Subjects will be randomized to a group who will be using the EWIS set infusion system for the initial Phase. All patients will be trained on the use of the EWIS infusion set by site staff and will be asked to demonstrate proficiency. All subjects will be instructed to change sets every 7 days or at set failure (replace with another Quick-set). At day 28 or after using 4 sets (set used defined as a set that was used for more than 6 hours), the patients will return to a visit, return all the extracted catheters sets and will switch to the Quickset infusion set, entering Phase 2. All patients will then be retrained on the use of the Quickset infusion set by site staff and demonstrate proficiency. After 28 days or after using 4 sets, the patients will all the extracted catheters sets .

An extension phase for additional one month (4 sets) will be conducted as a single arm to assess the seven day durability of sets.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes for at least one year
2. Using a MiniMed™ VEO pump or 640G Insulin pump with or without using an Enlite™ Sensor .
3. Age 18 to 80 years
4. Hemoglobin A1c level less than or equal to 10%
5. Not currently known to be pregnant, nor planning pregnancy during the study.
6. Willingness to follow the protocol and sign the informed consent

Exclusion Criteria:

1. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.
2. Pregnant or lactating females

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Primary | 8 weeks
  • Percent of catheters reaching 4, 5, 6, 7 days use without set failure.

SECONDARY OUTCOMES:
Exploratory outcomes | 8 weeks
  * Exploratory investigation of correlation between glycemia as measured by CGM records and pressure measurements, as recorded by the insulin pump.
  * Descriptive of site reactions. Pain at the infusion site device related issues (leakage, occlusion in fluid path, etc.).
  * Descriptive of set failure cases: accidental pull out, adhesive tape issues, infection, erythema and/or induration.
  * Descriptive of catheter explants:
    * Gross examination for cannula kinking and crimping.

OTHER OUTCOMES:
Adverse Events | 8 weeks
  * Diabetic ketoacidosis (DKA)
  * Severe hypoglycemia
  * Severe hyperglycemia
  * Serious adverse events (SAEs)
  * Unanticipated adverse device effects (UADEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No